CLINICAL TRIAL: NCT04655417
Title: is Ultrasound-guided Foam Sclerotherapy a Cost-effective Alternate for Treatment of Varicose Veins?
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Dr Anum Arif, Dr Anum Arif, Combined Military Hospital, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMHL
Record Dates: First submitted 2020-11-13; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Pain; Leg Edema; Cost Effectiveness; Cosmesis
MeSH Terms: conditions — Pain | interventions — Sodium Tetradecyl Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INTERVENTION GROUP (Experimental): SINGLE ARM OF PATIENTS WHO WILL RECEIVE SAME TREATMENT
  Interventions: Drug: Sodium Tetradecyl Sulfate

INTERVENTIONS:
Drug: Sodium Tetradecyl Sulfate — DRUG WILL BE INJECTED TO ALLAPTIENTS ACCORDING TO STANDARD PROTOCOL
  Other Names: STS

SUMMARY:
. It is the aim of this paper is to discuss our experience of foam sclerotherapy for varicose veins atour hospital

DETAILED DESCRIPTION:
we will manage all patients with vericose veins with injection sclerotherapy and will monitor there response in terms of relive in vsisble veins, swelling and pain.

we also want to evaluate hoe many sessions of injection sclerotherapy are required for complete resolution of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who present with symptomatic varicose veins underwent a duplex scan by radiologist to identify site of reflux and condition of deep veins. If the patient is a candidate for intervention then he is offered surgery or foam sclerotherapy

Exclusion Criteria:

* recurrent and secondary varicose veins

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-02-21 (Estimated); Study Completion 2021-02-21 (Estimated)

PRIMARY OUTCOMES:
pain by VAS score | 1 MONTH
  pain by VAS score
leg edema | 1 MONTH
  leg edema
cosmesis | 1 MONTH
  cosmesis
cost effectiveness | 1 MONTH
  cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Anum Arif, Principal Investigator — Combined military hospital lahore
Locations (1):
- Anum Arif, Lahore, Select A State Or Province, Pakistan

IPD SHARING:
Plan to Share IPD: No